CLINICAL TRIAL: NCT06538727
Title: A Feasibility and Pilot Study of an MRI Study to Investigate Changes After Osteopathic Manipulation Therapy in Patients With Myofascial Pain Syndrome
Brief Title: Pilot MRI Study on Osteopathic Manipulation for Myofascial Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Auburn University MRI Research Center (Unknown); Edward Via College of Osteopathic Medicine-Auburn (Unknown)
Responsible Party: Principal Investigator, Pao-Feng Tsai, Professor & Associate Dean for Research, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MPS2024
Record Dates: First submitted 2024-05-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial Pain; MPS; Myofascial Pain Syndrome; Myofascial Trigger Point
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: To achieve both aims, a two-arm-experimental design with a posttest control-group-only, will be conducted in a convenience sample of 20 adult patients with MPS of the upper back. Participants will be randomly allocated to one of the following three groups with a 1:1 ratio:
  * Group 1: receives one session of OMT
  * Group 2: control group - does not receive intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - One session of OMT Intervention (Experimental): Participants in the experimental condition will have one OMT treatment (Scapular Release) done to the upper back.
  Interventions: Other: Osteopathic Manipulation Treatment - Scapular Release
- Group 2 - No intervention (No Intervention): Participants in the control condition will receive no treatment.

INTERVENTIONS:
Other: Osteopathic Manipulation Treatment - Scapular Release — First, the patient will be positioned in the supine position. The physician or trained fellow will then place his/her hands on the medial border of the scapula on the affected side. From the paraspinal fascia to the medial border of the scapula a lateral traction is added along with a superior to inferior traction and additionally an inferior to superior traction. The shoulder will be used as an additional fulcrum by having the shoulder in the forward flexion position at 90 degrees and then adduction of the humerus to aid in addition movement of the scapula by moving the upper arm into adduction and abduction in a rhythmic motion. The treatment with a rhythmic and/or static traction in the motions described above and manual movement of the scapula will be done for a maximum of 15 minutes.
  Arms: Group 1 - One session of OMT Intervention

SUMMARY:
The goal of this clinical trial is to conduct MRI studies on adults with myofascial pain syndrome (MPS) to identify important MRI biomarkers that respond to OMT (osteopathic manipulation therapy) and investigate the feasibility of implementing MRI study and OMT in this population. The main outcomes of the study include:

* Determine whether biomarkers measured by MRI can differentiate normal tissues and MTrP (myofascial trigger point).
* Test the responsiveness of the biomarkers identified by MRI to the proposed intervention, OMT, in patients with MPS of the upper back.

Researchers will compare participants who will receive one session of OMT (Group 1 - Experimental Condition) and participants who will not receive any treatment (Group 2 - Control Condition) to see how the MRI-identified biomarkers respond to the intervention.

Participants will complete the following:

* Clinical screening
* MRI measures
* Battery of self-report surveys
* Clinical/Physical Function Assessment

DETAILED DESCRIPTION:
The goal of this clinical trial is to conduct MRI studies on adults with myofascial pain syndrome (MPS) to identify important MRI biomarkers that respond to OMT and investigate the feasibility of implementing MRI studies and OMT in this population. The main outcomes of the study include:

* Determine whether biomarkers measured by MRI can differentiate normal tissues and MTrP.
* Test the responsiveness of the biomarkers identified by MRI to the proposed intervention, OMT, in patients with MPS of the upper back.

Researchers will compare participants who will receive one session of OMT (Group 1 - Experimental Condition) and participants who will not receive any treatment (Group 2 - Control Condition) to see how the MRI identified biomarkers respond to the intervention.

Participants will complete the following tasks in the order below depending on their group assignment:

Experimental Group (Receives OMT Intervention):

* MRI pre-screening
* Clinical Screening:

  o Clinical assessment for identifying normal and MTrP tissues by a physician via palpation and verified by ultrasound imaging.
* Battery of self-report surveys

  * Pain Intensity Scale (PEG)
  * Pain Interference Scale (PEG)
  * Physical Function/Quality of Life Scale (PROMIS Physical Functioning Short Form 6B)
  * Sleep Scale (PROMIS Sleep Disturbance 6a+ Sleep Duration Question)
  * Pain Catastrophizing Scale (Pain Catastrophizing Scale - Short Form 6 item version)
  * Depression Scale (PHQ-9)
  * Anxiety Scale(GAD-7)
  * Global Satisfaction with Treatment Scale (PGIC)
  * Substance Abuse Screener (TAPS1).
  * Medication Intake Form
* Physical Function Assessment

  * Pain-Pressure Threshold measure (PPT)
  * Active Range of Motion measure (AROM)
  * Visual Analog Scale (VAS)
  * Neck Disability Index (NDI)
  * Sit to Stand Test (STS)
  * Get up and Go Test (GUG)
  * Six Minute Walk Test
* 1 hour of MRI Scans

  * Structural MRI
  * Diffusion Tensor MRI
  * fMRI (functional magnetic resonance imaging)
* Receive OMT Intervention (15-minute scapular release procedure)
* 1 hour of MRI Scans

  * Structural MRI
  * Diffusion Tensor MRI
  * fMRI
* Physical Function Assessment

  * Pain-Pressure Threshold measure (PPT)
  * Active Range of Motion measure (AROM)
  * Visual Analog Scale (VAS)

Control Group (No Intervention):

* MRI pre-screening
* Clinical Screening:

  o Clinical assessment for identifying normal and MTrP tissues by a physician via palpation and verified by ultrasound imaging.
* 1 hour of MRI Scans

  * Structural MRI
  * Diffusion Tensor MRI
  * fMRI
* Battery of self-report surveys

  * Pain Intensity Scale (PEG)
  * Pain Interference Scale (PEG)
  * Physical Function/Quality of Life Scale (PROMIS Physical Functioning Short Form 6B)
  * Sleep Scale (PROMIS Sleep Disturbance 6a+ Sleep Duration Question)
  * Pain Catastrophizing Scale (Pain Catastrophizing Scale - Short Form 6 item version)
  * Depression Scale (PHQ-9)
  * Anxiety Scale(GAD-7)
  * Global Satisfaction with Treatment Scale (PGIC)
  * Substance Abuse Screener (TAPS1).
  * Medication Intake Form
* Clinical/Physical Function Assessment

  * Pain-Pressure Threshold measure (PPT)
  * Active Range of Motion measure (AROM)
  * Visual Analog Scale (VAS)
  * Neck Disability Index (NDI)
  * Sit to Stand Test (STS)
  * Get up and Go Test (GUG)
  * Six Minute Walk Test

ELIGIBILITY:
Inclusion Criteria:

* MPS of the upper back with MTrPs as specified by Travell and Simons, with the confirmation of ultrasound procedure.
* Normal neurological examination including manual muscle testing, sensory exam, and deep tendon reflexes.
* English-speaking.
* Age 18 - 64 and reside in the community.

Exclusion Criteria:

* Malignancy.
* Major psychiatric disorders, such as bipolar disorder and depression.
* Cognitive impairment
* Skin lesion(s) on the shoulders and upper back.
* Systematic pain condition, such as Fibromyalgia.
* Previous surgical procedures in the spine, shoulder, and/or back within six months.
* Pregnancy.
* BMI of 40 or higher.
* Any health conditions that prevent participants from performing the experimental procedure
* Any contraindications of MRI procedure such as implantable cardiac devices (pacemakers, defibrillator, etc.), aneurysm clips, or metallic shoulder and/or spinal cord implants or screws.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
MRI Biomarkers - Structural MRI | For experimental group (Group 1): Outcomes will be assessed at Time 1 and Time 2 within the 4 hour duration; For no intervention group (Group 2): Outcomes will be assessed at Time 1 within the 4 hour duration.
  3D T1- weighted images (TR (repetition time) = 7 ms, TE (echo time) = 2.4 ms, resolution 0.6 mm3, flip angle = 20°, bandwidth = 790 Hz/pixel) will be used for high-resolution structural imaging. T2 maps will be obtained with T2 prepared gradient-echo (GRE) sequence with centric ordered k- space trajectory. T2 preparation duration will be varied from 24 ms to 84 ms in increments of 10 ms with sequence TR (time between consecutive T2 preps) = 3000 ms. The GRE acquisition parameters will be TR = 7 ms, flip angle = 6° (small flip angle to minimize T1 weighting), and resolution 0.6 mm 3 . T2 and proton density maps will be computed by voxel-wise non-linear fitting to mono-exponential T2 decay.
MRI Biomarkers - Diffusion Tensor MRI (DTI) | For experimental group (Group 1): Outcomes will be assessed at Time 1 and Time 2 within the 4 hour duration; For no intervention group (Group 2): Outcomes will be assessed at Time 1 within the 4 hour duration.
  The DTI will be acquired with a spin echo EPI (echo-planar imaging) sequence, at the same location as anatomical and T2 images, with TE/TR = 55/6000 msec, 2 mm3 isotropic resolution, BW (bandwidth) = 925 Hz/pixel, 12 gradient encoding directions, and b-values of 500 and 800 s/mm2. A Nonlinear least-squares fit will be used to determine the diffusion tensor out of the 12 diffusion weighted images according to the relationship as described before.
fMRI | For experimental group (Group 1): Outcomes will be assessed at Time 1 and Time 2 within the 4 hour duration; For no intervention group (Group 2): Outcomes will be assessed at Time 1 within the 4 hour duration.
  While all other measurements will be from the myofascial unit or region, fMRI will be acquired from the brain using a 2D gradient-echo multiband EPI (echo-planar imaging) sequence with TR = 1000 ms, TE = 20 ms, flip angle = 70°, voxel dimensions = 2 mm3 , and a multiband factor of 2. After standard pre-processing, brain activity and connectivity in the pain matrix will be assessed.

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) Assessment | For experimental group (Group 1): Outcomes will be assessed at Time 1 and Time 2 within the 4 hour duration; For no intervention group (Group 2): Outcomes will be assessed at Time 1 within the 4 hour duration.
  A research team member will use an algometer device to measure pressure pain threshold for each MTrP site and a normal tissue site on the opposite side of the upper back. The team member will measure each site for a total of three times, and these three measurements will be averaged for each MTrP site. The algometer will measure in lbs/in2.
Active Range of Motion (AROM) Assessment | For experimental group (Group 1): Outcomes will be assessed at Time 1 and Time 2 within the 4 hour duration; For no intervention group (Group 2): Outcomes will be assessed at Time 1 within the 4 hour duration.
  A goniometer will be used to measure in degrees, the participant's active range of motion. The neck, shoulder, forearm, and back will all be assessed. A separate range of motion in degrees based on the goniometer will be recorded for each body part.
Verbal Pain Report (VAS) Measure | For experimental group (Group 1): Outcomes will be assessed at Time 1 and Time 2 within the 4 hour duration; For no intervention group (Group 2): Outcomes will be assessed at Time 1 within the 4 hour duration.
  Participants will rate on a scale of 0-10 (Visual Analog Scale) how much pain they are currently experiencing in their upper back.
Neck Disability Index (NDI) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Measure self-report neck disability
Sit to Stand Test (STS) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Objective physical function measure
Get up and Go Test (GUG) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Objective physical function measure
Six Minute Walk Test | Outcome will be assessed at Time 1 within the 4 hour duration.
  Objective physical function measure
Pain Intensity Scale (PEG) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Pain
Pain Interference Scale (PEG) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Pain
Physical Function/Quality of Life Scale (PROMIS Physical Functioning Short Form 6B) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Physical function
Sleep Scale (PROMIS Sleep Disturbance 6a+ Sleep Duration Question) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Sleep
Pain Catastrophizing Scale (Pain Catastrophizing Scale - Short Form 6 item version) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Pain catastrophizing
Depression Scale (PHQ-9) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Depression
Anxiety Scale(GAD-7) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Anxiety
Global Satisfaction with Treatment Scale (PGIC) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Global satisfaction
Substance Abuse Screener (TAPS1) | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Substance abuse
Medication Intake Form | Outcome will be assessed at Time 1 within the 4 hour duration.
  Self-report survey-Medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Feng Tsai, PhD, Principal Investigator — Auburn University

IPD SHARING:
Plan to Share IPD: No